CLINICAL TRIAL: NCT05071209
Title: A Phase 1/ 2 Study of BAY 1895344 (Elimusertib, NSC#810486) in Pediatric Patients With Relapsed or Refractory Solid Tumors
Brief Title: Elimusertib for the Treatment of Relapsed or Refractory Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-10751; NCI-2021-10751 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PEPN2112 (Other: Pediatric Early Phase Clinical Trial Network); PEPN2112 (Other: CTEP); UM1CA228823 (NIH)
Record Dates: First submitted 2021-10-07; First posted 2021-10-08 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Alveolar Rhabdomyosarcoma; Recurrent Ewing Sarcoma; Recurrent Lymphoma; Recurrent Malignant Solid Neoplasm; Refractory Alveolar Rhabdomyosarcoma; Refractory Ewing Sarcoma; Refractory Lymphoma; Refractory Malignant Solid Neoplasm
MeSH Terms: conditions — Rhabdomyosarcoma, Alveolar; Sarcoma, Ewing; Lymphoma | interventions — BAY 1895344

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (elimusertib) (Experimental): Patients receive elimusertib PO BID on days 1-3, 8-10, 15-17, and 22-24 of each cycle. Treatment repeats every 28 days for 26 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Elimusertib

INTERVENTIONS:
Drug: Elimusertib — Given PO
  Other Names: ATR Inhibitor BAY1895344; ATR Kinase Inhibitor BAY1895344; BAY 1895344; BAY-1895344; BAY1895344

SUMMARY:
This phase I/II trial tests the safety, best dose, and whether elimusertib works in treating patients with solid tumors that have come back (relapsed) or does not respond to treatment (refractory). Elimusertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of BAY 1895344 (elimusertib) administered as an oral tablet, twice per day for 3 days on and 4 days off to patients < 18 years of age with recurrent or refractory Ewing sarcoma (and EWS fusions), PAX3-FOXO1 alveolar rhabdomyosarcoma, and non-central nervous system (CNS) solid tumors or lymphoma with specific deleterious deoxyribonucleic acid (DNA) damage response (DDR) pathway alterations. (Phase 1/Part A) II. To define the antitumor activity of BAY 1895344 (elimusertib) in pediatric patients and young adults with recurrent or refractory Ewing sarcoma (and EWS fusions). (Phase 2/Part B) III. To define the antitumor activity of BAY 1895344 (elimusertib) in pediatric patients and young adults with recurrent or refractory PAX3-FOXO1 fusion positive alveolar rhabdomyosarcoma. (Phase 2/Part B) IV. To define and describe the toxicities of BAY 1895344 (elimusertib) administered on this schedule. (Phase 1/Part A)

SECONDARY OBJECTIVES:

I. To characterize the pharmacokinetics of BAY 1895344 (elimusertib) in children and adolescents with recurrent or refractory cancer.

II. To assess the biologic activity of BAY 1895344 (elimusertib) by immunohistochemical assessments of phosphorylated (p)ATR, pH2AX, and pKAP1 in paired tissue samples before and after treatment with BAY 1895344 (elimusertib).

III. To assess whether the activity of BAY 1895344 (elimusertib) is influenced by alternative lengthening of telomeres (ALT), as well as tumor tissue expression of ATM, PGBD5, and/or R-loops.

IV. To assess whether the activity of BAY 1895344 (elimusertib) is associated with tumor mutational processes, as measured by whole genome tumor tissue sequencing.

V. To preliminary determine the anti-tumor activity of BAY 1895344 (elimusertib) in children < 18 years of age within the confines of a phase 1 study (Phase 1 and 2/Part A and B).

VI. To assess the antitumor activity of BAY 1895344 (elimusertib) in pediatric patients with non-CNS solid tumors or lymphomas with specific deleterious alterations in DDR pathway genes. (Phase 2/Part B)

OUTLINE: This is pediatric a phase I, dose-escalation study as well as a phase II dose expansion study in pediatric patients and young adults.

Patients receive elimusertib orally (PO) twice daily (BID) on days 1-3, 8-10, 15-17, and 22-24 of each cycle. Treatment repeats every 28 days for 26 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 12 months, every 6 months for 24 months, and then annually for up to 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Part A: Patients between >= 12 months and < 18 years of age
* Part B:

  * Patients between >= 12 months and =< 30 years of age for the phase 2 expansion cohorts for both EWS and PAX3-FOXO1 ARMS.
  * Patients between >= 12 months and =< 21 years of age for the phase 2 DDR expansion cohort

    * The Phase 2 cohorts will initially open concurrently with the Phase 1 portion but will only enroll patients at least 18 years of age. Patients < 18 years of age will be included in the Phase 2 cohorts only after the RP2D/MTD has been estimated in the Phase 1 portion
* All patients for both Parts A and B must have a minimum body surface area (BSA) >= 0.74 m^2
* All patients for both Parts A and B must have the ability to swallow BAY 1895344 (elimusertib) tablets intact
* Patients with recurrent or refractory solid tumors. Patients must have had histologic verification of malignancy at original diagnosis or relapse
* Part A: Any (non-CNS primary) solid tumor diagnosis including lymphoma which meets one of the following criteria:

  * Any Ewing Sarcoma (histological confirmation alone is adequate) or any EWS-fusion positive solid tumor (i.e. including related Ewing's family of tumors with EWS fusions such as EWS-WT1, EWS-ATF1, etc.)
  * Alveolar rhabdomyosarcoma (ARMS) with the PAX3-FOXO1 fusion. This does not include PAX7-FOXO1 or other variant fusion ARMS. Please note that a FISH showing FOXO1 breakapart is NOT sufficient for eligibility onto this cohort since it cannot distinguish between FOXO1 partners
  * Any (non-CNS primary) solid tumor including lymphoma with inactivating alterations of any of the DNA Damage Repair (DDR) genes: ATM, ATRX, BRCA1, BRCA2, CDK12, CHEK1, CHEK2, FANCA, MSH2, MRE11, PALB2, PARP1, POLD1, RAD51, or XRCC2
* Part B: Any (non-CNS primary) solid tumor diagnosis including lymphoma which meets one of the following criteria:

  * B1, EWS Cohort:

    * Any Ewing Sarcoma (histological confirmation alone is adequate) or any EWS-fusion positive solid tumor (i.e. including related Ewing's family of tumors with EWS fusions such as EWS-WT1, EWS-ATF1, etc.)
  * B2, PAX3-FOXO1 ARMS Cohort:

    * Alveolar rhabdomyosarcoma (ARMS) with the PAX3-FOXO1 fusion. This does not include PAX7-FOXO1 or other variant fusion ARMS. Please note that a FISH showing FOXO1 breakapart is NOT sufficient for eligibility onto this cohort since it cannot distinguish between FOXO1 partners
  * B3, DDR Non-statistical Cohort:

    * Any (non-CNS primary) solid tumor including lymphoma with inactivating alterations of any of the DNA Damage Repair (DDR) genes: ATM, ATRX, BRCA1, BRCA2, CDK12, CHEK1, CHEK2, FANCA, MSH2, MRE11, PALB2, PARP1, POLD1, RAD51, or XRCC2
* All the genes on the DDR panel are annotated with OncoKB, a precision oncology knowledge base which is publicly available here: https://www.oncokb.org/. Alterations which are categorized either 'Oncogenic' or 'Likely Oncogenic' would be considered sufficient for eligibility on either the phase 1 or phase 2 portions of this study. Alterations which are not annotated in OncoKB will need to be reviewed with locally qualified experts in molecular pathology, such as via an established molecular tumor board, in order to determine the likely oncogenicity AND will require approval by the study chair, Dr. Michael Ortiz. If such experts are not available at any institution, the study chair will review
* In cases where multiple mutations are present or multiple samples are available, either at different locations or different points in time, the presence of a single qualifying genomic alteration in any of those samples will is considered sufficient for eligibility on the phase 2 portions of this study
* Qualifying aberrations must be detected in either DNA or ribonucleic acid (RNA) in any tumor tissue sample (i.e. detection of a variant on circulating tumor DNA/RNA is not sufficient to qualify) using a somatic (and/or germline) mutational testing approach with either a targeted panel or whole exome/genome sequencing in the context of a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory setting. Any CLIA certified laboratory is acceptable to use
* Part A: Patients must have either measurable or evaluable disease
* Part B (1, 2, 3): Patients must have measurable disease
* Patients with a prior history of CNS metastases may enroll on study provided there is no current evidence of active disease at the time of enrollment
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2. Use Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50% for patients =< 16 years of age. Note that neurologic deficits in patients with tumors previously metastatic to the CNS (or other non-oncologic reasons) must have been stable for at least 7 days prior to study enrollment. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment. If after the required timeframe, the numerical eligibility criteria are met, e.g., blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive: >= 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Anti-cancer agents not known to be myelosuppressive (e.g., not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days after the last dose of agent
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Corticosteroids: If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g., pegfilgrastim) or 7 days for short acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell Infusions (with or without total-body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusions (DLI) or boost infusion: >= 84 days after infusion and no evidence of graft versus host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: >= 30 days
  * Cellular therapy: >= 42 days after the completion of any type of cellular therapy (e.g., modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * Radiation therapy (XRT)/external beam irradiation including protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow (BM) radiation
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131I MIBG): >= 42 days after systemically administered radiopharmaceutical therapy
  * Study specific prior therapy: Patients must not have received prior exposure to BAY 1895344 (elimusertib) or any other specific ATR inhibitors including berzosertib (M6620, VX-970), ceralasertib (AZD6738), M4344 (VX-803), M1774, and RP-3500. Treatment with other DNA damage repair inhibitors which do not specifically inhibit ATR (e.g. PARP inhibitors, WEE1 inhibitors, CHEK1 inhibitors, etc.) does not exclude them from eligibility on this study
* For patients with solid tumors without known bone marrow involvement

  * Peripheral absolute neutrophil count (ANC) >= 1000/uL
* For patients with solid tumors without known bone marrow involvement

  * Platelet count >= 100,000/uL (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* For patients with solid tumors without known bone marrow involvement

  * Hemoglobin >= 8.0 g/dL at baseline (may receive red blood cell [RBC] transfusions)
* Patients with known or possible bone marrow metastatic disease will be eligible for study provided they meet the blood counts in above inclusion criteria (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions). These patients will not be evaluable for hematologic toxicity. At least 5 of every cohort of 6 patients must be evaluable for hematologic toxicity for the dose-escalation part of the study. If dose-limiting hematologic toxicity is observed, all subsequent patients enrolled must be evaluable for hematologic toxicity
* Serum creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a creatinine based on age/gender as follows:

  * Age: 1 to < 2 years; Maximum serum creatinine (mg/dL): 0.6 (male); 0.6 (female)
  * Age: 2 to < 6 years; Maximum serum creatinine (mg/dL): 0.8 (male); 0.8 (female)
  * Age: 6 to < 10 years; Maximum serum creatinine (mg/dL): 1 (male); 1 (female)
  * Age: 10 to < 13 years; Maximum serum creatinine (mg/dL): 1.2 (male); 1.2 (female)
  * Age: 13 to < 16 years; Maximum serum creatinine (mg/dL): 1.5 (male); 1.4 (female)
  * Age: >= 16 years; Maximum serum creatinine (mg/dL): 1.7 (male); 1.4 (female)
* Bilirubin (sum of conjugated + unconjugated or total) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L. For the purpose of this study, the ULN for SGPT is 45 U/L
* Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled as evidenced by no increase in seizure frequency in the prior 7 days. For patients a history of seizure but not on anticonvulsants, no seizure in the past 3 months
* Nervous system disorders (Common Terminology Criteria for Adverse Events [CTCAE] version [v]5) resulting from prior therapy must be =< grade 2, with the exception of decreased tendon reflex (DTR). Any grade of DTR is eligible

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies, OR because there is yet no available information regarding human fetal or teratogenic toxicities. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use two effective methods of birth control, including a medically accepted barrier or contraceptive method (e.g., male or female condom) for the duration of the study and for 3 months + 2 days for males and 6 months + 2 days for females after receiving the last dose of BAY 1895344 (elimusertib) on the study. Abstinence is an acceptable method of birth control. Female patients must not breastfeed during treatment and until 4 months after last study drug administration
* Corticosteroids: Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible. If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients who are currently receiving drugs that are strong inducers or inhibitors of CYP3A4 are not eligible. Strong inducers or inhibitors of CYP3A4 should be avoided from 14 days prior to enrollment to the end of the study. Drugs that are considered sensitive or narrow therapeutic range CYP3A4 substrates should be avoided for the duration of protocol therapy
* Dedicated CNS imaging is not required but patients with current active CNS metastasis whether symptomatic or discovered incidentally without clinical symptoms, will be excluded from study participation
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 12 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Ortiz, Principal Investigator — Pediatric Early Phase Clinical Trial Network
Locations (29):
- United States (28):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
- Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1- Part A/ Dose Level 1; Phase 1- Part PK/ Dose Level 1: Patients with any Ewing Sarcoma or related EWS fusion, Alveolar rhabdomyosarcoma (ARMS) with the PAX3-FOXO1 fusion, or any (non- CNS primary) solid tumor. Patients < 18 years of age receive elimusertib 24 mg/m²/dose PO BID (maximum 40 mg/dose BID)
- Phase 2- Part B1/ Dose Level 1: Patients with any Ewing Sarcoma or any EWS-fusion positive solid tumor. Patients <18 years of age receive elimusertib 24 mg/m²/dose PO BID (maximum 40 mg/dose BID). Patients ≥ 18 years of age receive elimusertib 40 mg/dose PO BID
- Phase 2- Part B2/ Dose Level 1: Patients with PAX3-FOXO1 Alveolar Rhabdomyosarcoma (ARMS). Patients <18 years of age receive elimusertib 24 mg/m²/dose PO BID (maximum 40 mg/dose BID). Patients ≥ 18 years of age receive elimusertib 40 mg/dose PO BID
- Phase 2- Part B3/ Dose Level 1: Patients with any (non-CNS primary) solid tumor including lymphoma with inactivating alterations of any of the DNA Damage Repair (DDR) genes: ATM, ATRX, BRCA1, BRCA2, CDK12, CHEK1, CHEK2, FANCA, MSH2, MRE11, PALB2, PARP1, POLD1, RAD51, or XRCC2. Patients <18 years of age receive elimusertib 24 mg/m²/dose PO BID (maximum 40 mg/dose BID). Patients ≥ 18 years of age receive elimusertib 40 mg/dose PO BID
Period: Overall Study
Arm/Group | Phase 1- Part A/ Dose Level 1 | Phase 1- Part PK/ Dose Level 1 | Phase 2- Part B1/ Dose Level 1 | Phase 2- Part B2/ Dose Level 1 | Phase 2- Part B3/ Dose Level 1
Started | 8 | 1 | 10 | 9 | 3
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 1 | 10 | 9 | 3
Not completed — Lack of Efficacy | 8 | 1 | 9 | 8 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1- Part A/ Dose Level 1 | Phase 1- Part PK/ Dose Level 1 | Phase 2- Part B1/ Dose Level 1 | Phase 2- Part B2/ Dose Level 1 | Phase 2- Part B3/ Dose Level 1 | Total
Number analyzed (Participants) | 8 | 1 | 10 | 9 | 3 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 1 | 1 | 3 | 2 | 15
  Between 18 and 65 years | 0 | 0 | 9 | 6 | 1 | 16
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 13 [10 to 17] | 11 [11 to 11] | 20 [18 to 28] | 22 [14 to 26] | 18 [16 to 19] | 19 [10 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 6 | 8 | 1 | 20
  Male | 4 | 0 | 4 | 1 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2 | 1 | 1 | 6
  Not Hispanic or Latino | 6 | 0 | 8 | 8 | 2 | 24
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1
  White | 5 | 0 | 9 | 7 | 3 | 24
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 1 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Cycle 1 Dose Limiting Toxicities for BAY 1895344 (Elimusertib) During Dose Escalation
Description: Frequency (%) of patients experiencing a cycle 1 dose limiting toxicity among toxicity-evaluable patients stratified by dose level during the dose escalation part of the study (Part A).
Time Frame: Up to 28 days (cycle 1)
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1-Part PK/ Dose Level 1: Patients with any Ewing Sarcoma or related EWS fusion, Alveolar rhabdomyosarcoma (ARMS) with the PAX3-FOXO1 fusion, or any (non- CNS primary) solid tumor. Patients < 18 years of age receive elimusertib 24 mg/m²/dose PO BID (maximum 40 mg/dose BID)
Arm/Group | Phase 1- Part A/ Dose Level 1 | Phase 1-Part PK/ Dose Level 1
Number analyzed (Participants) | 8 | 1
Participants | 0 | 0

2. Primary Outcome: Response of BAY 1895344 (Elimusertib)
Description: Frequency (%) of patients with best response of complete response or partial response among response-evaluable patients stratified by Phase 2 cohort.
Time Frame: Through study completion, up to 37 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2- Part B1/ Dose Level 1 | Phase 2- Part B2/ Dose Level 1 | Phase 2- Part B3/ Dose Level 1
Number analyzed (Participants) | 10 | 9 | 3
Participants | 0 | 0 | 0

3. Secondary Outcome: Incidence of Adverse Events of BAY 1895344 (Elimusertib)
Description: Frequency (%) of patients with adverse events stratified by study part and dose level.
Time Frame: Through study completion, up to 37 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1- Part A/ Dose Level 1 | Phase 1- Part PK/ Dose Level 1 | Phase 2- Part B1/ Dose Level 1 | Phase 2- Part B2/ Dose Level 1 | Phase 2- Part B3/ Dose Level 1
Number analyzed (Participants) | 8 | 1 | 10 | 9 | 3
Participants | 8 | 1 | 8 | 9 | 3

4. Secondary Outcome: Area Under the Drug Concentration Time Curve of BAY 1895344 (Elimusertib)
Description: Median (min, max) of the area under the drug concentration time curve (AUC) in cycle 1 stratified by study part and dose level.
Time Frame: Up to 28 days
Population: Plasma concentrations were not collected for Part B patients as it was optional
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Phase 1- Part A/ Dose Level 1 | Phase 1- Part PK/ Dose Level 1
Number analyzed (Participants) | 8 | 1
hr*ng/mL | 7617 [3260.0 to 8354.0] | 7527 [7527.0 to 7527.0]

5. Secondary Outcome: Change in Phosphorylated (p)ATR of BAY 1895344 (Elimusertib)
Description: Median (min, max) of the change in (p)ATR stratified by study part and dose level.
Time Frame: Up to 28 days
Population: These were tissue-based assays to be performed on paired tissue samples, if available. There was no protocol mandated on study biopsy; tissue was to be available only when obtained for clinical purposes. No on-study tissue was obtained, submitted and available for this analysis
Arm/Group | Phase 1- Part A/ Dose Level 1 | Phase 1- Part PK/ Dose Level 1 | Phase 2- Part B1/ Dose Level 1 | Phase 2- Part B2/ Dose Level 1 | Phase 2- Part B3/ Dose Level 1
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Change in pH2AX of BAY 1895344 (Elimusertib)
Description: Median (min, max) of the change in pH2AX stratified by study part and dose level.
Time Frame: Up to 28 days
Population: as for outcome 5
Arm/Group | Phase 1- Part A/ Dose Level 1 | Phase 1- Part PK/ Dose Level 1 | Phase 2- Part B1/ Dose Level 1 | Phase 2- Part B2/ Dose Level 1 | Phase 2- Part B3/ Dose Level 1
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Change in pKAP1 of BAY 1895344 (Elimusertib)
Description: Median (min, max) of the change in pKAP1 stratified by study part and dose level.
Time Frame: Up to 28 days
Population: as for outcome 5
Arm/Group | Phase 1- Part A/ Dose Level 1 | Phase 1- Part PK/ Dose Level 1 | Phase 2- Part B1/ Dose Level 1 | Phase 2- Part B2/ Dose Level 1 | Phase 2- Part B3/ Dose Level 1
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Influence of ALT on Activity of BAY 1895344
Description: Median (min, max) of ALT in responders (CR or PR) versus non-responders among all response-evaluable patients.
Time Frame: Up to 28 days
Reporting Status: Not Posted

9. Secondary Outcome: Influence of Tumor Tissue Expression of ATM on Activity of BAY 1895344
Description: Median (min, max) of ATM in responders (CR or PR) versus non-responders among all response-evaluable patients.
Time Frame: Up to 28 days
Reporting Status: Not Posted

10. Secondary Outcome: Influence of Tumor Tissue Expression of PGBD5 on Activity of BAY 1895344
Description: Median (min, max) of PGBD5 in responders (CR or PR) versus non-responders among all response-evaluable patients.
Time Frame: Up to 28 days
Reporting Status: Not Posted

11. Secondary Outcome: Influence of Tumor Tissue Expression of R-loops on Activity of BAY 1895344
Description: Median (min, max) of R-loops in responders (CR or PR) versus non-responders among all response-evaluable patients.
Time Frame: Up to 28 days
Reporting Status: Not Posted

12. Secondary Outcome: Response of BAY 1895344 (Elimusertib) in Children < 18 Years
Description: Frequency (%) of patients with best response of complete response or partial response among response-evaluable patients in the dose escalation part of the study (Part A).
Time Frame: Up to 60 months
Reporting Status: Not Posted

13. Secondary Outcome: Response of BAY 1895344 in Pediatric Patients With Non-CNS Solid Tumors or Lymphomas
Description: Frequency of patients with best response of complete response or partial response among response-evaluable patients with non-CNS solid tumors or lymphomas with specific deleterious alternations in DDR pathway.
Time Frame: Up to 60 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through study completion, up to 37 months
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Phase 1- Part A/ Dose Level 1 | Phase 1- Part PK/ Dose Level 1 | Phase 2- Part B1/ Dose Level 1 | Phase 2- Part B2/ Dose Level 1 | Phase 2- Part B3/ Dose Level 1
All-Cause Mortality (participants affected / at risk) | 6/8 | 1/1 | 9/10 | 8/9 | 2/3
Serious Adverse Events (participants affected / at risk) | 7/8 | 1/1 | 8/10 | 9/9 | 3/3
Other Adverse Events (participants affected / at risk) | 8/8 | 1/1 | 10/10 | 9/9 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1- Part A/ Dose Level 1 (N=8) | Phase 1- Part PK/ Dose Level 1 (N=1) | Phase 2- Part B1/ Dose Level 1 (N=10) | Phase 2- Part B2/ Dose Level 1 (N=9) | Phase 2- Part B3/ Dose Level 1 (N=3)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 0 | 5 | 1 | 3
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Cardiac disorders - Other, Left atrial thrombus (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Extraocular muscle paresis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 4 | 0 | 4 | 6 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 3 | 0 | 3 | 2 | 2
Non-cardiac chest pain (General disorders and administration site conditions) | 0 | 0 | 1 | 2 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 0
Recurrent laryngeal nerve palsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
White blood cell decreased (Investigations) | 1 | 1 | 2 | 3 | 2
proptosis (Eye disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1- Part A/ Dose Level 1 (N=8) | Phase 1- Part PK/ Dose Level 1 (N=1) | Phase 2- Part B1/ Dose Level 1 (N=10) | Phase 2- Part B2/ Dose Level 1 (N=9) | Phase 2- Part B3/ Dose Level 1 (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 2 | 2 | 1
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0
Anemia (Blood and lymphatic system disorders) | 8 | 1 | 10 | 9 | 3
Anorexia (Metabolism and nutrition disorders) | 4 | 0 | 3 | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 5 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 3 | 3 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 4 | 5 | 0
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 1 | 0
Blurred vision (Eye disorders) | 1 | 0 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Cardiac disorders - Other, POTS (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Chloride Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Conduction disorder (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 3 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 | 1 | 0
Creatinine increased (Investigations) | 2 | 1 | 1 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 3 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 0 | 5 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0
Edema limbs (General disorders and administration site conditions) | 0 | 0 | 0 | 1 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 0 | 0 | 0 | 0
Eye disorders - Other, Puffiness below L eye (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, Type 1 Duane retraction syndrome (Eye disorders) | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0
Facial pain (General disorders and administration site conditions) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders and administration site conditions) | 2 | 1 | 6 | 4 | 2
Fever (General disorders and administration site conditions) | 0 | 1 | 2 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Gait disturbance (General disorders and administration site conditions) | 1 | 0 | 0 | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0
Gastrointestinal disorders - Other, Abdominal Cramping (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal disorders - Other, cyclical vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorders - Other, gastroparesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorders - Other, irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
General disorders and administration site conditions - Other, Chest tightness (General disorders and administration site conditions) | 0 | 0 | 1 | 0 | 0
General disorders and administration site conditions - Other, lightheadedness (General disorders and administration site conditions) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 7 | 2 | 3
Hematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Hepatobiliary disorders - Other, Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 3 | 0 | 5 | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 4 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2 | 3
Hypotension (Vascular disorders) | 3 | 0 | 4 | 4 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 2 | 0 | 0
Investigations - Other, Chloride Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Investigations - Other, Ferritin (Investigations) | 1 | 0 | 0 | 0 | 0
Irregular menstruation (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Left sided spontaneous 'twinge' of pain in ribcage, self resolves, Intermittent (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Localized edema (General disorders and administration site conditions) | 0 | 0 | 1 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 4 | 1 | 3 | 5 | 1
Malaise (General disorders and administration site conditions) | 0 | 0 | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, Ehlers-Danlos syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, Joint rang of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 0 | 4 | 7 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Nervous system disorders - Other, tremors (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 1 | 6 | 3 | 2
Non-cardiac chest pain (General disorders and administration site conditions) | 2 | 0 | 3 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders and administration site conditions) | 0 | 0 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 2
Pallor (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 3 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 2 | 1 | 8 | 6 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Psychiatric disorders - Other, Obsessive-compulsive disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Psychiatric disorders - Other, Panic attacks (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Psychiatric disorders - Other, Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Psychiatric disorders - Other, migraine with aura (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Psychiatric disorders - Other, non epileptic seizure (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Psychosis (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0
Renal and urinary disorders - Other, nocturnal enuresis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Reproductive system and breast disorders - Other, primary ovarian insufficiency (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, Restriction defect (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Right ventricular filling impaired (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 5 | 1 | 6 | 2 | 1
Skin and subcutaneous tissue disorders - Other, Keratosis pilaris (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, Skin hyperpigmentation (midback) (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urine discoloration (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Vaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 1 | 2 | 3 | 3
Weight gain (Investigations) | 0 | 0 | 1 | 0 | 0
Weight loss (Investigations) | 3 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
White blood cell decreased (Investigations) | 7 | 0 | 9 | 6 | 3
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
abdominal blister noted next to PleurX dressing - healing (Infections and infestations) | 1 | 0 | 0 | 0 | 0
blood draining w/pleural fluid (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
intermittent fatigue (General disorders and administration site conditions) | 1 | 0 | 0 | 0 | 0
intermittent hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
lightheadedness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
mononucleosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
mouth swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
numbnuess noted above umbilicus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
pruritic rash on forearm d/t bandage sensitivity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
ptosis left eye (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
teeth feel "loose" (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT05071209/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT05071209/ICF_001.pdf